CLINICAL TRIAL: NCT04007874
Title: Open-label Randomized Controlled Trial for the Effects of Continuous Ethinylestradiol/Levonorgestrel (30/150 μg/Day) Compared With Vitamin E (400 IU/Day) in the Treatment of Menstrually-related Migraine and Migraine During Perimenopause
Brief Title: Oral Contraceptive Pill Compared With Vitamin E in Women With Migraine
Acronym: WHATT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Netherlands Brain Foundation (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, G.M. Terwindt, MD, Head of headache clinic, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WHATT; 2018-004096-12 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Migraine; Migraine;Menstrual
Keywords: Migraine; Women; Hormones; Oral contraceptive pill; Vitamin E
MeSH Terms: conditions — Migraine Disorders | interventions — Ethinyl Estradiol; Levonorgestrel; Vitamin E

STUDY DESIGN:
Intervention Model Description: Open-label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ethinylestradiol/levonorgestrel (Experimental): Ethinylestradiol/levonorgestrel 30/150 µg oral tablets once daily without a stopweek for 3 months
  Interventions: Drug: Ethinylestradiol/levonorgestrel
- Vitamin E (Active Comparator): Vitamin E 400 IU oral capsules once daily for 3 months
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Ethinylestradiol/levonorgestrel — Ethinylestradiol/levonorgestrel 30/150 µg oral tablets once daily without a stopweek for 3 months
  Other Names: Microgynon 30; RVG 08204
  Arms: Ethinylestradiol/levonorgestrel
Drug: Vitamin E — Vitamin E 400 IU oral capsules once daily for 3 months
  Arms: Vitamin E

SUMMARY:
Open-label randomized controlled trial to study the efficacy of continuous daily use of ethinylestradiol/levonorgestrel (30/150 µg/day) compared with vitamin E (400 IU/day) in the treatment of women with menstrually-related and perimenopausal migraine.

DETAILED DESCRIPTION:
Rationale: The prevalence of migraine is three times higher in women than in men. Clinical and epidemiological studies suggest a prominent role for sex hormones in female migraine patients. Menstruation is an important factor increasing the susceptibility for an upcoming attack. Perimenstrual migraine attacks are also more disabling, longer lasting, and more difficult to treat than other attacks. Hormonal fluctuations during menopausal transition are associated with increased susceptibility for migraine as well, whereas hormonal changes in migraine during pregnancy seem to be associated with decreased attack frequency. Thus, sex hormonal conditions seem to affect the susceptibility for migraine attacks in women, but there is a lack of understanding the underlying pathophysiological mechanism. Currently, there is no clear evidence-based hormonal intervention for the treatment of migraine in women. The investigators hypothesize that continuous daily use of an oral contraceptive pill will be an effective, well-tolerated preventive treatment for 1) menstrually-related migraine and 2) perimenopausal migraine.

Objective: To study the efficacy of continuous daily use of ethinylestradiol/levonorgestrel (30/150 µg/day) compared with vitamin E (400 IU/day) in the treatment of menstrually-related and perimenopausal migraine.

Study design: Open-label randomized controlled trial. Study population: Women with menstrually-related or pure menstrual migraine and women with perimenopausal migraine.

Intervention: Continuous daily use of ethinylestradiol/levonorgestrel (30/150 µg/day) compared with vitamin E (400 IU/day).

Primary endpoint: Change in monthly migraine days from baseline to the last 4 weeks of treatment (weeks 9-12).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study will encompass a period of 4 months (1 baseline month and 3 treatment months). Patients have to fill out daily headache diaries throughout the study using a web-based app (≈ 5 min). Patients visit the headache clinic thrice, once for inclusion, once during the baseline period and once after 3 months of therapy (duration ≈ 1 hour). During the first and last visit blood samples will be taken. Patients will be contacted twice during follow-up to evaluate (S)AE's. Treatment with the oral contraceptive pill is accompanied by a very low risk of developing thromboembolisms. Participation might benefit participants by reducing their migraine attack frequency or intensity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Premenopausal with menstrual migraine OR migraine during the early menopausal transition phase (a difference of 7 days or more in length of consecutive cycles, which should occur at least twice in a period of 12 menstrual cycles)
* Demonstrated at least 80% compliance with eDiary during baseline period
* No or stable for at least two months on prophylactic medication

Exclusion Criteria:

* Smoking
* Migraine with aura
* Chronic migraine with 15 or more headache days per month/with 8 or more migraine days per month
* Medication-overuse headache (ICHD-3 criteria)
* Women who are breastfeeding, pregnant, or planning to become pregnant
* Oral contraceptive use and not willing to undergo washout period (stop for two consecutive months)
* Vitamin E use at start of the study
* Use of other sex hormone containing treatments
* Increased risk of VTE: history of VTE or thrombophlebitis, hereditary predisposition for VTE (APC resistance, protein C or S deficiency, antithrombin deficiency), VTE in first-degree family member at young age, long term immobilisation
* Increased risk of ATE: history of ATE, hereditary predisposition for ATE (hyperhomocysteinemia, antiphospholipid antibodies), ATE in first-degree family member at young age, diabetes mellitus, total cholesterol ≥ 6.5
* Other contraindication for oral contraceptives: liver malignancy, schistosomiasis, HIV/aids, use of immunosuppressives, tuberculosis, sex-hormone-dependent malignancies (breast, endometrial or ovary carcinomas), pancreatitis, vaginal bleeding with unknown cause, other diseases that can influence vessels (malignancies, heart valve disorders, atrial fibrillation, SLE, haemolytic uremic syndrome, chronic inflammatory bowel disease, sickle cell disease)
* Contraindication for vitamin E: vitamin K deficiency
* Hypersensitivity for any of the compounds in oral contraceptive or vitamin E
* Spontaneous postmenopausal status (menstrual bleedings have ceased for 12 consecutive months)
* Iatrogenic postmenopausal status
* Inability to complete the electronic diary in an accurate manner
* Any serious illness that can compromise study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of migraine days | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in monthly migraine days

SECONDARY OUTCOMES:
Number of headache days | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in monthly headache days
Number of migraine attacks | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in monthly migraine attacks
Number of probable migraine attacks | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in monthly probable migraine attacks
Number of 50% responders | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Patients who had ≥50% reduction in the number of migraine days
(Serious) adverse events | Up to 3 months
  Occurrence of adverse events and serious adverse events

OTHER OUTCOMES:
Number of 75% responders | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Patients who had ≥75% reduction in the number of migraine days
Number of complete responders | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Patients who had 100% reduction in the number of migraine days
Number of acute treatment days | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in monthly acute treatment days
Mean migraine severity score/day | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in migraine severity (four-point anchored scales (0=none, 1=mild, 2=moderate, and 3=severe))
Mean migraine-related symptom severity score/day | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in migraine-related symptom severity (four-point anchored scales (0=none, 1=mild, 2=moderate, and 3=severe))
Migraine-Specific Quality of life questionnaire (MSQ) | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in Migraine-Specific Quality of life questionnaire (MSQ) total score (range from 14 (mild impact) to 84 (severe impact))
Headache Impact Test (HIT-6) | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in Headache Impact Test (HIT-6) total score (range between 36 (mild impact) - 78 (severe impact))
Perceived Stress Scale (PSS) | From baseline to the last 4 weeks of treatment (weeks 9-12)
  Change in Perceived Stress Scale (PSS) total score (range between 0 (mildly stressed) - 40 (severely stressed))

CONTACTS AND LOCATIONS:
Overall Officials: Gisela M Terwindt, MD,PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Arend BWH, van Casteren DS, Verhagen IE, MaassenVanDenBrink A, Terwindt GM. Continuous combined oral contraceptive use versus vitamin E in the treatment of menstrual migraine: rationale and protocol of a randomized controlled trial (WHAT!). Trials. 2024 Feb 15;25(1):123. doi: 10.1186/s13063-024-07955-8. PMID 38360739